CLINICAL TRIAL: NCT03754231
Title: Validation Study on RENEW's Aingeal at KK Women's and Children's Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Renew Group (Industry)
Responsible Party: Principal Investigator, Low Bao Bei Kelly, Associate Consultant, Department of Paediatrics, KK Women's and Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/2223 (Paediatric)
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Vital Sign; Heart Rate; Respiratory Rate
Keywords: Vital sign monitoring; Heart rate; Respiratory rate

STUDY DESIGN:
Intervention Model Description: All patients recruited will be wearing the Aingeal device at a paediatric outpatient clinic setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aingeal (Experimental): All recruited patients will wear the Aingeal device as a form of heart rate monitoring and respiratory rate monitoring in a paediatric outpatient clinic setting.
  Interventions: Other: Heart rate monitoring; Other: Respiratory rate monitoring

INTERVENTIONS:
Other: Heart rate monitoring — The heart rate of recruited patients will be monitored for 15 minutes over 2 phases:
  i) 10 minutes at rest ii) 5 minutes during physical activity in the form of walking or playing
Other: Respiratory rate monitoring — The heart rate of recruited patients will be monitored for 15 minutes over 2 phases:
  i) 10 minutes at rest ii) 5 minutes during physical activity in the form of walking or playing

SUMMARY:
This proposal describes the evaluation of a CE-marked, FDA cleared vital signs Surveillance Monitoring system in a paediatric outpatient population in KK Women's and Children's Hospital ("KKH"), the main tertiary women and children hospital in Singapore. User acceptance of Aingeal and the Surveillance System will be considered within the clinical settings.

DETAILED DESCRIPTION:
RENEW's Surveillance Monitoring system is made up of two main components:

a patient-worn wireless vital signs monitor (Aingeal) that transmits data over Wi-Fi to a central station software platform (Surveillance Station). The Aingeal device measures single lead ECG, heart rate, respiration waveform and rate, and skin temperature. A snapshot of data is transmitted by the devices intermittently to the Surveillance Station, enabling vital signs trends to be plotted. This proposal describes the evaluation of RENEW's Aingeal device in a paediatric outpatient population in KK Women's and Children's Hospital ("KKH"), the main tertiary women and children hospital in Singapore. In the paediatric population, assessment of RENEW's Aingeal device will include the accuracy of the device at deriving heart rate from single lead ECG and at deriving respiratory rate when compared against a commonly used vital signs monitor. User acceptance of Aingeal and the Surveillance System will be considered within the clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Male or female paediatric patients, aged between 3 and 17 years
* Patients attending outpatient care at KK Women's and Children's Hospital, Singapore

Exclusion Criteria:

* Patients with active, implantable devices (such as a pacemaker or ICD)
* Patients with any skin condition or injury affecting the electrode placement site
* Patients that are pregnant
* Those patients who, in the opinion of the clinic staff, are not suitable to participate.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Heart rate comparison | 15 minutes
  Heart rate is calculated manually via ECG waveform and compared against the Aingeal device using Bland Altman approach

SECONDARY OUTCOMES:
Respiratory rate comparison | 15 minutes
  Repiratory rate measurement is compared between Aingeal device and Capnostream device using Bland Altman approach.

CONTACTS AND LOCATIONS:
Overall Officials: Bao Bei Kelly Low, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT03754231/Prot_SAP_000.pdf